CLINICAL TRIAL: NCT00730951
Title: The Evaluation and Standardization of Ginseng and Its Components for Blood Pressure Regulation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Unity Health Toronto (Other)
Collaborators: Heart and Stroke Foundation of Ontario (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 107460
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Asian ginseng; Starch

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): 0.5g Korean Red Ginseng (1 capsule) 5.5g Corn Starch (11 capsules)
  Interventions: Dietary Supplement: Korean Red Ginseng; Dietary Supplement: Corn Starch
- 2 (Experimental): 1g Korean Red Ginseng (2 capsules) 5g Corn Starch (10 capsules)
  Interventions: Dietary Supplement: Korean Red Ginseng; Dietary Supplement: Corn Starch
- 3 (Experimental): 3g Korean Red Ginseng (6 capsules) 3g Corn Starch (6 capsules)
  Interventions: Dietary Supplement: Korean Red Ginseng; Dietary Supplement: Corn Starch
- 4 (Experimental): 6g Korean Red Ginseng (12 capsules)
  Interventions: Dietary Supplement: Korean Red Ginseng
- 5 (Experimental): 6g Corn Starch Control (12 capsules)
  Interventions: Dietary Supplement: Corn Starch

INTERVENTIONS:
Dietary Supplement: Korean Red Ginseng — 500mg Capsulated Ground Dried Korean Red Ginseng Root
  Arms: 1; 2; 3; 4
Dietary Supplement: Corn Starch — 500mg Capsulated Corn Starch
  Arms: 1; 2; 3; 5

SUMMARY:
While the use of herbals is increasing considerably, their efficacy and safety in the humans remains largely unknown. This surge in demand prompts a call for its evaluation. Preliminary data demonstrates that KRG can affect vascular function and our research group has previously shown that Korean Red Ginseng (KRG) can lower blood pressure (BP) in hypertensive individuals. However, it is unknown which dose is the most effective in producing a desired effect. To address this issue, we will test escalating doses of a single Korean red ginseng batch of 0.5g, 1g 3g and 6g on BP in patients with hypertension to determine the most efficacious dose. The most promising dose will be extracted and will advance to next level to be tested again on BP control. The findings of the study may result in better ginseng standardization.

DETAILED DESCRIPTION:
Individuals will arrive at the Risk Factor Modification Centre, St. Michael's Hospital between the hours of 8:00 and 10:00am after a 10 to 12-hour fast on seven separate mornings. They will not have consumed any antihypertensive medications on the study mornings. Each visit will be separated by a minimum of a week. Since the half-life of ginsenosides in humans is less than 24-hours, to allow for a washout of approximately seven half-lives.

In each of the four studies, when individuals arrive at our clinic on a test day they will first have their weight measured and subsequently rest in the seated position. They will then have a catheter inserted into a forearm vein, which will be kept patent by saline. From this device, a registered intravenous nurse will obtain a series of 7ml blood samples. Blood will be taken at 30-min intervals. Subsequently, individuals will fill out forms detailing their pharmacological regimen for the previous 24-hours and their diet (dinner) and activity (sleep, urination, morning routine) regimen for the previous 12-hours. As well, they will detail any adverse events that they experienced since their previous visit. Individuals will then have their office BP measured with a mercury sphygmomanometer until three consecutive measurements of both SBP and DBP <5 mmHg different are obtained. At this point, BP should be steady and subjects will be fitted with an ABPM. Measurements will be taken every 5-min for 30-min, for a total of seven measurements. After the seventh measurement (time 0-min), measurements will be taken automatically every 10-min for 180-min. At time 0-min, treatment or placebo capsules will be consumed. At time 60-min a 360-calorie Ensure® breakfast will be consumed within 5-min. Blood samples will be drawn at 30-min intervals, starting at time 0-min. For 24-hours after the ingestion of treatment, a record of any side effects will be detailed by the participants and then provided to us.

ELIGIBILITY:
Inclusion Criteria:

* Essential Hypertension

Exclusion Criteria:

* Secondary Hypertension
* Diabetes
* Chronic Kidney Disease
* Liver Disease
* Unstable Angina
* Coronary / Cerebrovascular event in the previous 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2007-06; Primary Completion 2008-01 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Blood Pressure will be measured with an Ambulatory Blood Pressure Monitor | every 5 min for first 30 min, then every 10 minutes for 180 minutes

SECONDARY OUTCOMES:
Blood samples will be drawn and tested for Nitric Oxide levels. | every 30 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Vladimir Vuksan, PhD, Principal Investigator — Clinical Nutritian and Risk Factor Modification Centre
Locations (1):
- Clinical Nutrition and Risk Factor Modification Centre, Toronto, Ontario, Canada